CLINICAL TRIAL: NCT07356492
Title: Expanding Veteran Sponsorship Initiative+ to Support High-Risk Transitioning Servicemembers and Veterans: A Precision Medicine Approach (PEC 24-113)
Brief Title: Expanding Veteran Sponsorship Initiative+ to Support High-Risk Transitioning Servicemembers and Veterans: A Precision Medicine Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VISN 2 Mental Illness Research, Education and Clinical Center (Unknown); VISN 17 Center of Excellence for Research on Returning War Veterans (Unknown); Department of War Study to Assess Risk & Resilience in Servicemembers - Longitudinal Study (Unknown); James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency); Health Economics Resource Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEX 25-001; 1I50HX003929-01 (Other Grant/Funding Number: VA ORD)
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Reintegration Difficulties; Suicidal Ideation and Behaviors; Health; Connectedness
Keywords: Suicide; Reintegration; Social Determinants of Health; Transitioning Servicemember/Veteran; Suicide Prevention; VA Utilization; Community Intervention; Suicidal Behavior
MeSH Terms: conditions — Suicidal Ideation; Behavior; Suicide; Suicide Prevention | interventions — Community Support

STUDY DESIGN:
Intervention Model Description: Methods: The purpose of this PEI proposal is to evaluate VSI expansion into VSI+ utilizing four III Armored Corps installations (FY2026-2027). The evaluators will use a pragmatic cluster-randomized trial design. This design will allow us to extend implementation support to the maximal number of military installations and enhance our formative evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Transition as Usual (No Intervention): Arm 1. Transition as Usual, n=900
  * receives no Onward Ops services
  * receives no VA stepped care services
- Veteran Sponsorship Initiative Base (Experimental): Arm 2. VSI Base, n=900
  * receives Onward Ops peer sponsor and community services
  * receives no VA stepped care services
  Interventions: Behavioral: Onward Ops- receive peer sponsor and community support
- Veteran Sponsorship Initiative+ (Experimental): Arm 3. VSI+, n=900
  * receives Onward Ops peer sponsor and community services
  * receives VA stepped care services
  Interventions: Behavioral: Onward Ops- receive peer sponsor and community support; Behavioral: VA stepped care services

INTERVENTIONS:
Behavioral: Onward Ops- receive peer sponsor and community support — Onward Ops is a nonprofit organization dedicated to supporting U.S. military service members and their families as they transition from active duty to civilian life. It provides a structured, community-based approach to help ease the challenges of reintegration. Participants may engage in either the Onward Ops Solo or Co-Op track. Both tracks provide access to the Onward Ops dashboard- an online platform to manage transition plans, track progress, and explore curated resources. In addition, Co-Op participants are matched to a community-based, peer sponsor & receive assistance from community partners.
  Other Names: ETS Sponsorship
  Arms: Veteran Sponsorship Initiative Base; Veteran Sponsorship Initiative+
Behavioral: VA stepped care services — The high-risk TSMVs receive approximately five sessions of VSI+ with optimally two sessions occurring prior to discharge with a TRICARE approved referral. VSI+ is delivered via telehealth video to allow flexibility and to accommodate the fact that TSMVs will be moving after discharge. The topics and tasks associated with each session involve items such as confirming TSMVs completed their VHA registration and VBA service-connected disability application, made contact with their VSI sponsor, submitted their military records to enable them to receive a VHA eligibility group, and directly connecting TSMVs to VHA primary care. Because VSI+ is designed as an adjunctive service and TSMVs may require a broad range of services and resources, the VSI+ social workers ensure ongoing communication with VSI sponsors, community partners, VHA primary care and mental health providers. TSMVs will have seamless access to the NVCC with ability to receive primary and specialty care.
  Arms: Veteran Sponsorship Initiative+

SUMMARY:
Background Young Veterans in the U.S. face a heightened risk of suicide, particularly during the first year after leaving military service-a period often referred to as the "deadly gap." Suicide rates among Veterans aged 18 to 34 have nearly doubled since 2001, and research shows that reintegration challenges during this transition are closely linked to increased suicide risk.

The Veteran Sponsorship Initiative (VSI) was developed to address this critical period by connecting Transitioning Servicemembers and Veterans (TSMVs) with trained, VA-certified peer sponsors. These sponsors help TSMVs navigate civilian life and access VA care. Early evaluations show that TSMVs matched with sponsors are more likely to report lower levels of reintegration difficulties, higher levels of social support, engage in VA services and report lower rates of depression and suicide risk.

This project enhances VSI by integrating predictive analytics-developed in partnership with Harvard Medical School and the DoW STARRS-LS team-to identify high-risk TSMVs before they leave the military. Those identified receive not only a sponsor but also targeted VA mental and health care services. This hybrid effectiveness-implementation study will evaluate the impact of this enhanced model (VSI+) on mental health outcomes and VA engagement among 2,700 high-risk TSMVs.

Method/Design

The purpose of this PEI proposal is to evaluate VSI expansion into VSI+ with enrollment occurring on four US Army installations (FY2026-2027). The study employs a pragmatic cluster-randomized trial with embedded mixed-method implementation evaluation to compare three arms:

1. Transition as Usual (TAU)
2. VSI Base= peer sponsorship and community support
3. VSI+= VSI Base plus VA stepped care services

The evaluation is guided by the RE-AIM framework to assess:

* Reach (enrollment rates)
* Effectiveness (reintegration difficulties, depression, anxiety, suicidal ideation/behavior, and VA utilization outcomes)
* Adoption (site and staff uptake)
* Implementation (fidelity and feasibility)
* Maintenance (sustainability)

Study Aims

1. Effectiveness: Evaluate the impact of VSI Base and VSI+ on reintegration difficulties, depression, anxiety, suicidal ideation/behavior, and VA utilization outcomes.
2. Implementation: Assess the feasibility and fidelity of implementing VSI Base and VSI+ across multiple sites using a bundled strategy.
3. Economic Impact: Estimate the budget impact of VSI Base and VSI+ on healthcare costs, including inpatient, emergency, and outpatient care.

DETAILED DESCRIPTION:
Young Veterans in the U.S. are experiencing a suicide epidemic, with suicide rates for Veterans aged 18 to 34 years old more than doubling from 2001 (23.6 per 100,000) to 2021 (49.6 per 100,000; VA, 2023). In 2020, the rate of suicide among Veterans of this age group was 1.52 times higher than among older Veterans and 2.61 times higher than among same-aged non-Veterans (VA, 2022a). Notably, the risk for suicide is significantly elevated for young TSMVs during their transition from active-duty military service to civilian life. A VA Office of Mental Health and Suicide Prevention study showed that suicide rates after separation are time-dependent, with the highest suicide rates observed in the first year after discharge. These rates increased over the first 6 months and then generally peaked in the 6 to 12 months after discharge (Ravindran et al., 2020). Given the significant increase in suicide risk during this transitional period, researchers have dubbed the time between discharge and successful reintegration into civilian life as the "deadly gap" (Geraci et al., 2020a; Sokol et al., 2021) and have indicated that preventive interventions for this vulnerable population should begin prior to discharge (Vogt et al., 2020). About 200k TMSVs exit active-duty service yearly (VA, 2018).

To assist, the VSI is the first large-scale implementation of an evidence-based practice that intervenes with TSMVs prior to discharge. It attempts to reduce TSMV suicide risk by decreasing psychological pain often associated with the transition, increasing connectedness and assisting TSMVs to safely store their firearms by pairing of TSMVs with certified, volunteer, community-based sponsors (1-on-1). VSI is based on the DoW's Permanent Change of Station Sponsorship program and recommendations from the DoW's Best Practices Identified for Peer Support Programs (2011). On four III Armored Corps (US Army) military installations, TSMVs have had the opportunity, since FY2020 to complete a US Army Soldier for Life (SFL) application six months prior to their military discharge. SFL is a US Army program, separate from Army Transition Assistance Program, that facilitates access to services provided by the VA, local communities, and Veteran-friendly service organizations. When completing the SFL application, TSMVs have the option to request a VA VSI sponsor.

ETS Sponsorship (2025) is a national nonprofit organization that serves as the national operational partner for VSI, through its Onward Ops program, as part of a VA memorandum of agreement with the VHA Undersecretary for Health and is responsible for managing the process of collecting, securing and storing information provided by TSMVs from the SFL application. Within 14 days of completing the SFL application and requesting a sponsor, TSMVs participate in an intake with an Onward Ops transition coordinator to identify reintegration needs and then are matched with a best fitting sponsor based on geographical location, gender, sexual orientation, interests and desired profession. After matching, sponsors have regular contact with their TSMVs through social media, email, and monthly video or in-person meetings and help TSMVs to identify Specific-Measurable-Achievable-Relevant-Time Bound (SMART) goals related to domains of reintegration and social determinants of health (Geraci et al., 2020b). Contact continues through approximately 6 months post-discharge.

Sponsors are managed by different community partners (e.g., nonprofits, private hospitals, or county veteran service offices) across the country. These community partners are vetted by both the VA's National Center for Healthcare Advancement and Partnerships (2025) and Onward Ops. Primary responsibilities of the community partners include: (a) recruiting volunteer sponsors and ensuring they attend VA certification training (see Geraci et al., 2020b, for more information on the certification training); (b) matching TSMVs with sponsors; (c) managing sponsors' relationships with TSMVs in their local region; (d) submitting referrals to other agencies to assist TSMVs in meeting their goals and (e) accessing and monitoring TSMV progress in the initiative using a common digital dashboard, in partnership with Google Public Sector. Onward Ops attempts to balance the number of TSMVs in its program desiring a sponsor with the number of available sponsors and has shown an ability to recruit and certify the needed number of sponsors with many sponsors volunteering to work with more than one TSMV at a time.

In FY2022, VSI+ was developed by the VA Transitioning Servicemember/Veteran Suicide Prevention Center (TASC), housed at the James J. Peters VAMC and jointly supported by the VISN 2 MIRECC and VISN17 Center of Excellence. TASC, in partnership with Dr. Ronald Kessler, Dr. Brian Marx (VA National Center for PTSD) and the DoD STARRS team. VSI+ added a precision medicine approach to the original VSI, hereafter referred to as "VSI Base". The VSI+ has two key components:

The first component of VSI+ is screening TSMVs for suicide risk pre-discharge with the STARRS calculator (Kearns et al., 2023), which was developed using machine learning models that predicted post-discharge suicide attempt based on a constrained number of item-level, self-report survey predictors which are accessed in real-time by TASC to determine risk levels. The team found that 30% of Soldiers with the highest predicted risk on the final STARRS calculator included 92.5% of self-reported suicide attempts post-discharge. The resulting 17 predictors/questions in the calculator have already been added to the SFL application and completed by over 25,000 TSMVs since April 2023.

The second is VA Stepped-Care Intervention & Case Management. As detailed within the VA/DoD Clinical Practice Guideline for Assessment and Management of Patients at Risk for Suicide (VA/DoD, 2019), social work case management has been shown to decrease psychiatric readmission rates, decrease cost of care, and improve continuity of care for high-risk individuals. There are many case management interventions that already exist to reduce suicidal behaviors during periods of transition as well as to manage more general behavioral and psychosocial problems that occur during periods of transition (Yen et al., 2019). In VA, for example, an effective program exists in which peer specialists with a history of criminal justice involvement collaborate with VA social workers to provide case management for Veterans transitioning out of prison back to the community (Kim et al., 2019). As integrated into the current VSI+ manual developed by the TASC team, VSI+ social workers follow the professionally recognized and VHA-adopted framework for evidence-based case management practices (VA, 2019), with a sequential set of steps and associated tasks that consist of comprehensive assessment, need identification, problem solving and goal identification, planning and implementation, referrals and transition, monitoring and evaluation.

After receiving TSMV enrollment data, VA VSI+ social workers contact and invite high-risk TSMVs to participate in VSI+. The high-risk TSMVs receive approximately five sessions of VSI+ with optimally two sessions occurring prior to discharge with a TRICARE approved referral. VSI+ is delivered via telehealth video to allow flexibility and to accommodate the fact that TSMVs will be moving after discharge. The topics and tasks associated with each session involve items such as confirming TSMVs completed their VHA registration and VBA service-connected disability application, made contact with their VSI sponsor, submitted their military records to enable them to receive a VHA eligibility group, and directly connecting TSMVs to VHA primary care. Because VSI+ is designed as an adjunctive service and TSMVs may require a broad range of services and resources, the VSI+ social workers ensure ongoing communication with VSI sponsors, community partners, VHA primary care and mental health providers.

The VA National Virtual Care Clinic (NVCC) for Transitioning Veterans was established in 2022 by TASC/VSI teams to help the VA to provide timely and personalized access to critical VA care for TSMVs as soon as possible after discharge. Through a charter with the VHA Office of Primary Care, the VCC expanded to five regional hubs across the nation with the goal of providing virtual VA healthcare to TSMVs within 3 months of military discharge. Since its inception, the VCC has already conducted 4,000 encounters with TSMVs as it has addressed the primary care and additional needs identified during the primary care appointment, such as mental health, physical therapy, Whole Health, Women's Health and polytrauma/traumatic brain injury.

Methods: The purpose of this PEI proposal is to evaluate VSI expansion into VSI+ utilizing four III Armored Corps installations (FY2026-2027). The evaluators will use a hybrid type 2 effectiveness-implementation evaluation with a sequential roll-out to participating military installations over time to allow us to extend implementation support to the maximal number of military installations and enhance formative evaluation. The study employs a pragmatic cluster-randomized trial with embedded mixed-method implementation evaluation to compare three arms.

Participants (n=2,700) will be enrolled on military installations approximately six months prior to discharge and provide data at baseline (as part of the SFL application), six months after discharge (VA Qualtrics survey) and 12 months after discharge (Qualtrics). The investigators will conduct cluster-randomization based on two-week time intervals. The investigators will randomize two-week intervals ahead of time that will determine which high-risk Soldiers are enrolled within Arm 2 (VSI Base) vs. Arm 3 (VSI+) based on which time interval the Soldiers enroll. High risk TSMVs for the TAU arm will be identified through case-control matching using the Fuzzy Python procedure to match TSMVs in the VSI Base and VSI+ arms to 900 high risk TSMVs who opted to not receive an Onward Ops sponsor or other Onward Ops services.

Measures: Reintegration difficulties (Primary Outcome) will be broadly assessed during each timepoint using the Military to Civilian Questionnaire (M2C-Q; Sayer et al., 2011), a 16-item measure that assesses difficulties in (a) interpersonal relationships with family, friends, and peers; (b) productivity at work, school, or home; (c) community participation; (d) self-care; (e) leisure; and (f) perceived meaning in life. The Columbia-Suicide Severity Rating Scale (CSSRS) Screener (Bjureberg et al., 2021) will be administered during each timepoint based on the more comprehensive full-length version of the scale (Posner et al., 2011). The screener is designed to measure suicidal ideation severity and suicidal behaviors with two subsets of items. The Patient Health Questionnaire-2 (PHQ-2; Kroenke et al., 2003) is a measure of depression and will be administered at each timepoint. The Generalized Anxiety Disorder (GAD-2; Kroenke et al., 2007) is a measure of anxiety and will be administered at each timepoint. VA enrollment and utilization will also be measured.

Aim 1: VSI+ Effectiveness. The first aim is to further determine the effectiveness of VSI+, as evidenced by measures of reintegration difficulties, depression, anxiety, suicidal ideation/behaviors, and VA utilization with three arms (Arm 1. TAU, n=900; Arm 2. VSI Base, n=900; and Arm 3. VSI+, n=900). Consistent with CONSORT guidelines for 3-arm trials (Juszczak et al., 2019), the primary hypothesis is that TSMVs in VSI Base (Arm 2) and VSI+ (Arm 3), when the data from the separate arms is collapsed and combined, will experience less reintegration difficulties (primary outcome), less suicidal ideation/behaviors, less depression and improved VA utilization compared to TSMVs within the TAU. The secondary hypothesis is that TSMVs randomly assigned to VSI+ (Arm 3) will experience less reintegration difficulties, less suicidal ideation/behaviors, less depression, less anxiety, and improved VA utilization compared to VSI Base (Arm 2) TSMVs.

Aim 2: Implementation. The second aim is to determine the feasibility and potential utility of a stakeholder-engaged plan for implementing the VSI+ on four III Armored Corps installations. A phased, bundled implementation strategy was developed according to the QUERI Implementation Roadmap (Goodrich et al., 2020; Kilbourne 2019) and the Expert Recommendations for Implementing Change taxonomy (Powell et al., 2015) based on needs and barriers identified in earlier evaluations of VSI (Geraci et al., 2022). Strategies have been selected as appropriate to the unique challenges of implementation phase - pre-implementation, implementation, and sustainment. As a prerequisite to studying the implementation strategies empirically, the evaluators followed the reporting specifications provided by Proctor and colleagues (2013) specific to naming, clearly describing, and operationalizing the respective implementation strategies. The investigators anticipate that the implementation strategies will assist in addressing the following barriers: (a) perceived competing priorities by local VA and community partners; (b) lack of awareness of the initiative; (c) challenges of coordinating and communicating across many stakeholders (nonprofit; local, state and federal agencies); and (d) need for sustained funding.

Aim 3: Budget Impact Analysis of VSI Base and VSI+. The budget impact analysis will estimate the impact of adopting VSI+ compared to VSI-base and TAU related to health care costs. The investigators will follow the general recommendations from the International Society for Pharmacoeconomics and Outcomes Research (Sullivan et al., 2014) on conducting budget impact analysis. The investigators will conduct this analysis from the societal perspective and include VA-provided and VA-purchased health care costs, non-VA health care costs, and the costs of VSI Base and VSI+. The hypotheses are consistent to those within Aim 1 but specific to inpatient and emergency care costs and VERA generation. The investigators project that identified costs will be offset through VERA generation and less inpatient and emergency care costs for VSI-base and VSI+ participants.

Data Analysis: HLM8 (Raudenbush et al., 2019) will be used to create a hierarchical linear model for each outcome. Intent-to-treat analyses will be utilized. Time will be included as a Level 1 predictor as a linear pattern of change with a static time term for each time point. Time will be centered at Time-3 so that the parameter for the intercept will represent the outcomes at the 12 month assessment (O'Connor et al., 2014). The investigators will create the full model by including orthogonal contrasts at Level 2 to test the hypotheses. As described by CONSORT guidelines (Juszczak et al., 2019) and recommended by Feingold and colleagues (2013) for 3-arm trials, the first contrast will test the primary hypothesis of VSI Base (Arm 2=1/3) and VSI+ (Arm 3=1/3) vs. TAU (-2/3) and the second contrast will test the secondary hypothesis of VSI+ (Arm 3=.5) vs. VSI Base (Arm 2= -.5). Effect size will be calculated using procedures outlined by Feingold (2013).

Sample Size: The investigators calculated the sample size needed given the stepped-wedge design to test the primary hypothesis with the primary outcome variable. The calculations were based on having 80% power at a significance level of 0.05 to detect a medium effect size (partial eta of .06) between the arms on M2C-Q. The total number of TSMVs needed to be enrolled across the four military installations will be 420 per arm. This was determined after adjusting the total sample size required under randomization, for the design effect, and accounting for attrition between enrollment and the 12 month post-discharge assessment. The investigators are enrolling a larger sample than needed to facilitate analysis for the secondary variable, suicidal ideation/behavior. Based on the STARRS data (Kearns et al., 2023), the investigators anticipate that prevalence of suicidal behavior in the 12 months after separation will be 4% for STARRS high-risk TSMVs. The investigators plan to use a .05-level two-sided test to evaluate the intervention effect. If VSI+ is associated with a 50% reduction in risk, statistical power will be greater than 0.9 to detect this effect. If VSI+ is associated with a 33% reduction in risk, statistical power will be greater than 0.8. If VSI+ is associated with a 25% reduction in risk, statistical power will be 0.68.

ELIGIBILITY:
Inclusion Criteria:

* TSMVs must be 18-years of age or older
* Enroll prior to military discharge
* Be planning to transition from one of the target military installations' included in the evaluation during an active enrollment window

Exclusion Criteria:

* The participants Army STARRS score cannot identify the TSMV as low risk nor as acute high risk for suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Military to Civilian Questionnaire (M2C-Q; Sayer et al., 2011) | Change in baseline scores across 3 timepoints [Time frame: Baseline, 6 months post-military separation, and 12 months post-military separation]
  Reintegration difficulties will be assessed using the Military to Civilian Questionnaire (Primary Outcome; M2C-Q; Sayer et al., 2011), a 16-item measure that assesses reintegration difficulties in (a) interpersonal relationships with family, friends, and peers; (b) productivity at work, in school, or at home, (c) community participation; (d) self-care; (e) leisure, and (f) perceived meaning in life. Items are rated on a 5-point Likert scale ranging from 0 (No difficulty) to 4 (Extreme difficulty). Minimum: 0 (best); Maximum: 4 (worst)

SECONDARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS) screener (Posner et al., 2011) | Change in baseline scores across 2 timepoints [Time Frame: Baseline and 12 months after]
  Risk for suicidal ideation and behaviors will be assessed using procedures described by Katz et al. (2019). The VA Intake team will ask questions from the Columbia-Suicide Severity Rating Scale (C-SSRS) screener (Posner et al., 2011) supplemented by questions based on cues provided in the full C-SSRS about suicide attempts ("Have you attempted suicide or done harm to yourself or put yourself in a dangerous situation with the intent of ending your life"), and about injuries ("Did it result in you needing to get medical care with a doctor or hospital"). TSMVs will be placed in hierarchical categories based on their highest level of reported ideation or behavior. Minimum: 0 (best); Maximum: 7 (worst)
Patient Health Questionnaire-2 (PHQ-2; Kroenke et al., 2003) | Change in baseline scores across 3 timepoints [Time Frame: Baseline, 6 months after, and 12 months after]
  Depression will be assessed using the Patient Health Questionnaire-2 (PHQ-2; Kroenke et al., 2003), a 2-item self-report measure that has shown strong construct validity, test-retest reliability, and internal reliability across samples (Kroenke et al., 2003). A PHQ-2 score ranges from 0-6. If the score is 3 or greater, major depressive disorder is likely.
Generalized Anxiety Disorder-2 (GAD-2; Kroenke, K. et al., 2007). | Change in baseline scores across 3 timepoints [Time Frame: Baseline, 6 months after, and 12 months after]
  Anxiety will be assessed using the GAD-2, a 2-item self-report measure that has shown strong construct validity, test-retest reliability, and internal reliability across samples (Kroenke et al., 2007). A GAD-2 score ranges from 0-6. If the score is 3 or greater, an anxiety depressive disorder is likely.
VA Primary Care Utilization | Program entry through 12 months post-discharge of the last TSMV to enroll
  VA primary care utilization serves as a key indicator of access to and continuity of care, reflecting how effectively Veterans are connected to routine, preventive, and chronic disease management services. Higher or sustained primary care utilization is often associated with improved health outcomes, reduced emergency department visits, and better chronic disease management among Veterans. This will be assessed through the VA Corporate Data Warehouse (CDW), which enables us to access data for TSVMs who have enrolled and utilized VA healthcare services
VA healthcare enrollment and utilization | Program entry through 12 months post-discharge of the last TSMV to enroll
  VA healthcare enrollment and utilization will be assessed through the VA Corporate Data Warehouse (CDW), which enables us to access data for TSMVs who have enrolled and utilized VA healthcare services. Vanneman et al. (2015) conducted one of the first studies to identify predictors of VA enrollment and utilization for TSMVs. Importantly, they identified that there was a three-fold increase in VA enrollment and utilization during the first-year post-discharge for TSMVs who engaged in VA healthcare services prior to discharge. Therefore, this evaluation will begin the enrollment process early for TSMVs while they are still within the military.
Suicide attempt requiring medical care | Program entry through 12 months post-discharge of the last TSMV to enroll
  This measure captures incidents where a Veteran engages in a suicide attempt that results in the need for medical intervention, including emergency care, hospitalization, or other acute clinical services. It serves as a critical indicator of acute suicide risk and the effectiveness of prevention, intervention, and postvention strategies within the VA healthcare system. This will be assessed through the VA Corporate Data Warehouse (CDW), which enables us to access data for TSVMs who have enrolled and utilized VA healthcare services.
Reach | Program entry through 12 months post-discharge of the last TSMV to enroll
  Reach will be assessed by calculating the percent of eligible TSMVs that sign up for the Sponsorship Initiative compared to the total number of eligible TSMVs on respective military installations.
Adoption (Military Installation) | Program entry through 12 months post-discharge of the last TSMV to enroll
  Adoption will be assessed by the percent of military installations that continue through the study.
Adoption (VA Social Workers) | Program entry through 12 months post-discharge of the last TSMV to enroll
  Adoption will be assessed by the percent of VA social workers that continue through the study.
Maintenance (VA funding) | Time point: After implementation on the last Army installation
  Maintenance (VA funding) will be evaluated after the implementation phase and operationalized as the amount of funding dedicated to the sustainment and expansion of the sponsorship initiative.
Cost of Healthcare | Final evaluation at final timepoint [Time Frame: 12 months after last TSMV exists the military]
  We will conduct this analysis from the societal perspective and include VA-provided and VA-purchased health care costs, non-VA health care costs, and the costs of VSI Base and VSI+.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C Geraci, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center; Richard W Seim, Principal Investigator — Central Texas Veterans Health Care System Waco VA Medical Center, Waco, TX; Emily R Edwards, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center; Marianne S. Goodman, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center; Brigid B Connelly, MA, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO; Erin P Finley, PhD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Jean Yoon, PhD MHS, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA; David E Goodrich, EdD MS MA, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: VA Veteran Sponsorship Initiative — https://www.mirecc.va.gov/visn17/vsi.asp